CLINICAL TRIAL: NCT03598335
Title: Characterizing Malignant Tumors Using Ultrasound Doppler Imaging
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-0096-17
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Malignant Tumor of Women's Reproductive System
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Women with malignant tumor: Women with malignant tumor in reproductive system
  Interventions: Device: Ultrasound
- Women with benign tumor: Women with benign tumor in reproductive system
  Interventions: Device: Ultrasound
- Women with no observed tumor: Women with no observed tumor in reproductive system
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound imaging of women arriving at clinic for routine care

SUMMARY:
The aim of this study is to determine whether Ultrasound Doppler imaging can identify malignant tumors at a very early stage.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting for routine abdominal/vaginal ultrasound

Exclusion Criteria:

* Pregnant women

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women presenting at the Hillel Yaffe Medical Center gynecological ultrasound clinic.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Early characterization of malignant tumors | One year
  Comparison of Ultrasound Doppler findings at different speeds between women without tumors, with benign tumors and with malignant tumors of reproductive system

CONTACTS AND LOCATIONS:
Overall Officials: Alon Shrim, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel